CLINICAL TRIAL: NCT05044052
Title: Do Peer-comparisons, Emphasis on Harms, and/or Inclusion of Viral Prescription Pad Resources Increase Responsiveness to Feedback About Antibiotic Prescribing in Primary Care: Protocol for Two Linked Trials With Embedded Process Evaluations (OH Trial)
Brief Title: Does Inclusion of Viral Prescription Pad Resources Increase Responsiveness to Feedback About Antibiotic Prescribing in Primary Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Women's College Hospital (Other)
Collaborators: Ontario Agency for Health Protection and Promotion (Other Government); College of Family Physicians of Canada (Other); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Noah Ivers, Family Physician, Canada Research Chair (Tier 2) in Implementation of Evidence Based Practice, Women's College Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 2020-0024-E (OH Trial)
Record Dates: First submitted 2021-09-03; First posted 2021-09-14 (Actual); Last update posted 2023-01-05 (Actual); Status verified 2023-01

CONDITIONS: Infection
Keywords: audit and feedback; antibiotics
MeSH Terms: conditions — Infections

STUDY DESIGN:
Intervention Model Description: Cluster Randomized Control Trial
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group - Viral prescription pad + emphasis (Experimental): Physicians in this group will receive their usual MyPractice: Primary Care report from Ontario Health. This report will include antibiotic prescribing indicators as well as a link to the viral prescription pad. As part of the intervention, these physicians will also receive additional emphasis on the viral prescription pad by 1) encouraging it in the dissemination email of the MyPractice feedback report, and (2) mailing a paper version of the viral prescription pad with instructions on embedding the viral prescription pad into the recipient's EMR.
  Interventions: Behavioral: Emphasis on the Choosing Wisely Viral Prescription Pad
- Control group (No Intervention): Physicians in this group will receive their usual MyPractice: Primary Care report from Ontario Health. This report will include antibiotic prescribing indicators as well as a link to the viral prescription pad. This group will not receive any additional emphasis on the viral prescription pad and will not receive a paper copy in the mail.

INTERVENTIONS:
Behavioral: Emphasis on the Choosing Wisely Viral Prescription Pad — We will investigate the effects of emphasizing the use of materials developed by Choosing Wisely Canada (CWC) - namely the viral prescription pad - to help physicians act upon the feedback to reduce their prescribing.
  Arms: Intervention Group - Viral prescription pad + emphasis

SUMMARY:
Antibiotic overuse is common and antibiotic prescribing contributes to rising rates of antimicrobial resistance. Primary care physicians prescribe the majority of all antibiotics and there is large inter-physician variability in prescribing that cannot be explained by differences in patient populations.

In Ontario, audit and feedback (A&F) is routinely offered to primary care providers from a variety of sources. Ontario Health - an agency created by the Government of Ontario - provides A&F via email to physicians who voluntarily sign up for their "MyPractice" reports. These are multi-topic reports with aggregated (physician-level) data. As of November 2021, the MyPractice reports for family physicians will include data on antibiotic prescribing. To date, less than half of Ontario family physicians have signed up for the MyPractice reports from Ontario Health.

For this study, the investigators will conduct a trial to investigate the effect of adding viral prescription pad resources to family physician A&F received through a MyPractice: Primary Care report. This evaluation provides an opportunity to determine if the addition of this resource to an A&F intervention increases changes to antibiotic prescribing.

DETAILED DESCRIPTION:
This study will examine ways to optimize the effects of A&F for antibiotic prescribing in primary care. This study will aim to determine if emphasis (or not) on the use of a viral prescription pad developed by Choosing Wisely Canada (CWC) can help physicians act upon the feedback from their MyPractice report to reduce their antibiotic prescribing.

Antibiotic prescribing feedback within the multi-topic MyPractice: Primary Care report will be sent to family physicians who signed up for this program from Ontario Health. This report includes a link to the Choosing Wisely viral prescription pad. Physicians will be randomized to the control group or intervention group. Physicians in the intervention group will receive additional emphasis on the use of the viral prescription pad and will also have a paper copy of the prescription pad mailed to their practice.

One month after the initial intervention, participants will be invited to complete a process evaluation survey to determine why or why not the intervention worked and how individual factors can affect physician motivation, willingness, and ability to engage in new practices. Intervention participants will also be invited to take part in a process evaluation interview.

ELIGIBILITY:
Inclusion Criteria:

* Family physicians who sign up for the MyPractice reports by September 2021

Exclusion Criteria:

* Family physicians who did not sign up for the MyPractice reports by September 2021

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3379 (Actual)
Dates: Start 2021-12-15 (Actual); Primary Completion 2022-06-15 (Actual); Study Completion 2022-12-15 (Actual)

PRIMARY OUTCOMES:
Antibiotic prescribing rate | 6 months
  Total number of antibiotic prescriptions per 1000 65+ patient visits

SECONDARY OUTCOMES:
Proportion Antibiotic Rx with Prolonged Duration | 6 months
  Antibiotics prescribed for more than 7 days per episode
Proportion Antibiotic Rx with Prolonged Duration | 12 months
  Antibiotics prescribed for more than 7 days per episode
Antibiotic drug costs | 6 months
  Cost in CDN$
Antibiotic drug costs | 12 months
  Cost in CDN$
Antibiotics prescribed for viral infections | 6 months
  Total number of antibiotic rx per 1000 65+ patient visits for presumed viral condition (and thus likely unnecessary) based on administrative database diagnostic codes
Antibiotics prescribed for viral infections | 12 months
  Total number of antibiotic rx per 1000 65+ patient visits for presumed viral condition (and thus likely unnecessary) based on administrative database diagnostic codes
Total Antibiotic Days of Therapy | 6 months
  Total number DOTs per 1000 65+ patient visits
Total Antibiotic Days of Therapy | 12 months
  Total number DOTs per 1000 65+ patient visits
Proportion of broad spectrum antibiotic prescriptions | 6 months
  antibiotic prescriptions that are broad spectrum
Proportion of broad spectrum antibiotic prescriptions | 12 months
  antibiotic prescriptions that are broad spectrum

CONTACTS AND LOCATIONS:
Overall Officials: Noah M Ivers, MD, Principal Investigator — Women's College Hospital
Locations (1):
- Women's College Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
No plan to share this data

REFERENCES:
- [Derived] Shuldiner J, Lacroix M, Saragosa M, Reis C, Schwartz KL, Gushue S, Leung V, Grimshaw J, Silverman M, Thavorn K, Leis JA, Kidd M, Daneman N, Tradous M, Langford B, Morris AM, Lam J, Garber G, Brehaut J, Taljaard M, Greiver M, Ivers NM. Process evaluation of two large randomized controlled trials to understand factors influencing family physicians' use of antibiotic audit and feedback reports. Implement Sci. 2024 Sep 16;19(1):65. doi: 10.1186/s13012-024-01393-5. PMID 39285305
- [Derived] Shuldiner J, Schwartz KL, Langford BJ, Ivers NM; Ontario Healthcare Implementation Laboratory study team. Optimizing responsiveness to feedback about antibiotic prescribing in primary care: protocol for two interrelated randomized implementation trials with embedded process evaluations. Implement Sci. 2022 Feb 14;17(1):17. doi: 10.1186/s13012-022-01194-8. PMID 35164805